CLINICAL TRIAL: NCT01590940
Title: Use of Parietex Plug-and-patch Hernia Mesh in Elective Open Inguinal Hernia Repair: A Pilot Investigation
Brief Title: Use of Parietex Plug and Patch Hernia System in Open Inguinal Hernia Repair
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Owen Drive Surgical Clinic of Fayetteville (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: ODSC001
Record Dates: First submitted 2012-05-02; First posted 2012-05-03 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-05

CONDITIONS: Evaluate the Use of a New Mesh Type in Open Inguinal Hernia Repair
MeSH Terms: interventions — Melanocyte-Stimulating Hormones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Parietex mesh: Enrolled patients who met criteria for inclusion would have undergone open inguinal hernia repair using the Parietex plug and patch hernia system
  Interventions: Procedure: Open inguinal hernia repair with mesh

INTERVENTIONS:
Procedure: Open inguinal hernia repair with mesh

SUMMARY:
The use of synthetic mesh plugs for open inguinal hernia repair has seen dramatic variability in the number and composition of meshes currently on the world market. The use of biomaterials (PLLA, PGA) in hernia mesh is a relatively new and innovative method. These selected polymers have the ability to degrade while implanted, allowing for sufficient natural tissue healing and scarring. This usage presumably favors a decrease in foreignness, inflammatory reaction, recurrence, and incidence of chronic groin pain. Prior studies with similar plug meshes in the same indication have yielded favorable results which require this mesh to be investigated in its specific application.

Primary Objective

Evaluate the incidence of peri-operative and post-operative complications after the application of the Parietex plug and patch hernia system in open inguinal hernia repair. We will assess the efficacy of this mesh by examination and the application of a pain scale at the following intervals: 1 month, 3 months, and 1 year, respectively. Assessment is intended to evaluate:

* Patient report of pain via their Pain score
* Wound complication
* Incidence of chronic groin pain
* Recurrence rate
* Other complications Secondary Objectives

Record the description and assessment of the Parietex plug and patch hernia system:

* surgical technique
* description of dissection and mesh placement
* method of fixation
* operative times, anesthesia choice
* length of hospital stay
* mesh handling characteristics
* return to daily activities
* overall patient satisfaction

DETAILED DESCRIPTION:
This is a post-market single center pilot study to evaluate the efficacy and safety of the Parietex plug and patch hernia system following open inguinal hernia repair.

The Parietex plug and patch hernia system is composed of:

* a pre-cut patch made from lightweight monofilament polyester
* a semiresorbable disk which is a bio-component made of polyester monofilament and poly-L-lactic acid (PLLA).

Patients who meet criteria for the study will be invited to join the study at their consult prior to surgery. F. Andrew Morfesis M.D. FACS will consent the patient, and offer to answer questions and address concerns. Once the patient has provided informed consent, they will be given a hernia surgery specific survey (mesh specific quality of life scale) that will test parameters such as pain, discomfort in movements, and pain frequency. Post operatively, research assistants will review the chart to collect data on secondary objectives from the Operative Note. This data will be entered into a secure excel database.

It will be explained by Dr. Morfesis that these questionnaires must be completed in-person during subsequent follow-up visits. Follow-up visits will be scheduled at 1 month, 3 months, and 1 year, at which time the patient will be examined, and will fill out the hernia surgery specific measure to evaluate pain at follow up. If patients cannot be scheduled for their follow-up visits, pain questionnaires will be given over the phone by a research assistant to reduce data loss.

Subject Selection

This study will include 50 patients following the criteria described below:

Inclusion Criteria

* All patients regardless of gender > 18 years of age presenting with inguinal hernias.
* Subjects will be informed of the nature of the study, and have provided signed written consent.

Exclusion Criteria

Excluded groups will include:

* children under the age of 18
* subjects that meet criteria for biologic mesh placement
* emergency procedure
* recurrent hernias.

Withdrawal Criteria Subjects may withdraw or be withdrawn from the study at any time. The reason for discontinuation will be collected. Additionally, subjects may be withdrawn from the study by the principle investigator for noncompliance with study procedures.

Study Assessments

The study subjects will be evaluated at the following time points:

Screening (pre-operative) Patients will be informed by Dr. Morfesis about the nature of the study and if they are in agreement to participate the signed consent will be obtained.

Prior medical/surgical history will be obtained at time of consultation. Any additional testing or imaging that may be needed will also be obtained before the time of surgery.

Patients will receive a pre-operative hernia pain scale. This scale has been tailored after numerous validated hernia mesh scales assessing types of pain, frequency of pain, and quality of life.

Procedure OR time Intra-operative device related adverse events Technique Method of fixation Length of hospital stay Mesh handling Type of anesthesia

Follow-up will occur at 1 month, 3 months, and 1 year visit Patients will fill out the hernia pain scale. Wound examination Scar thickness and appearance Suture infections Post-operative device related adverse events Recurrence Chronic groin pain Other complications

ELIGIBILITY:
Inclusion Criteria:

* All patients regardless of gender > 18 years of age presenting with inguinal hernias.
* Subjects will be informed of the nature of the study, and have provided signed written consent.

Exclusion Criteria:

* children under the age of 18
* subjects that meet criteria for biologic mesh placement
* emergency procedure
* recurrent hernias.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: n=50 males and females age 18 and up
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Florias A Morfesis, M.D., Principal Investigator — Owen Drive Surgical Clinic; Brian P Rose, B.S., Study Chair — The Brody School of Medicine at East Carolina University
Locations (1):
- Owen Drive Surgical Clinic of Fayetteville, Fayetteville, North Carolina, United States